CLINICAL TRIAL: NCT01320631
Title: Male Sexual Experience and Its Impact on Quality of Life Before and After Their Sexual Partners Undergo Polypropylene Mesh Augmented Pelvic Floor Reconstruction
Acronym: SEXQ
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Other Study IDs: R09-08-008
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Sacral Colpopexy; Pelvic Organ Prolapse
Keywords: uterine prolapse; vaginal prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The correction of the pelvic organ protrusion is aimed at restoring the pelvic floor functional status and ultimately improving the patient's quality of life. There are a few studies that have explored the effect of pelvic reconstructive surgery on female sexual function (1,2) but no studies have evaluated the male partner's sexual experience. The investigators intend to use a newly psychometrically validated questionnaire to capture this aspect. The sexual experience questionnaire (SEX-Q) is the first questionnaire to solely and exclusively combine functional and quality of life concepts (erection, individual satisfaction, and couple satisfaction domains) in a brief questionnaire, which allows a more focused and less burdensome evaluation of the sexual experience in men (3). Another issue is the density of the mesh material and if it can be felt vaginally even if it is not eroded and to what degree this might bother the male partner during intercourse.

ELIGIBILITY:
Inclusion Criteria:

1. Sexually active couple at the time of pre-operative visit
2. Female partner scheduled to undergo a mesh augmented repair

Exclusion Criteria:

1. Not sexually active
2. Use of other graft material than polypropylene mesh
3. Contraindications to surgery based on existing medical conditions
4. Pregnancy
5. Desire for pregnancy in the future

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male sexual partners of women who are sexually active and are scheduled to undergo a mesh augmented repair for pelvic organ prolapse referred to the Division of Urogynecology and Reconstructive Pelvic Surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantic Health System, Morristown, New Jersey, United States

REFERENCES:
- [Derived] Culligan PJ, Haughey S, Lewis C, Priestley J, Salamon C. Sexual Satisfaction Changes Reported by Men After Their Partners' Robotic-Assisted Laparoscopic Sacrocolpopexies. Female Pelvic Med Reconstr Surg. 2019 Sep/Oct;25(5):365-368. doi: 10.1097/SPV.0000000000000574. PMID 29494351